CLINICAL TRIAL: NCT06991946
Title: Real-world Patient-centric Study to Assess the Feasibility of a Molecular Diagnosis on Treatment Decision Making for Patients With Metastatic Breast Cancer in Spain (HOPE-Focus)
Brief Title: Patient-Centric Study to Assess the Impact of Genomic Profiling on the Treatment of Patients With Metastatic Breast Cancer in Spain
Acronym: HOPE-Focus
Status: Recruiting | Type: Observational
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Roche Farma, S.A (Industry); Menarini Group (Industry); AstraZeneca (Industry); Pfizer (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: SOLTI-2401
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
Keywords: molecular advisory board; molecular tumor board; genomic data; targeted therapy; patient-centric trial; observational trial; Molecular data; genomic analysis; liquid biopsy; tumor block
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection and archival tumor tissue collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metastatic breast cancer of any subtype: Patients with metastatic breast cancer of any subtype that have progressed after at least one line of treatment in the metastatic setting
  Interventions: Genetic: Liquid Biopsy; Genetic: Archival Tumor DNA
- ER+/HER2- metastatic breast cancer: Patients recently diagnosed with ER+/HER2- metastatic breast cancer as a recurrence during adjuvant treatment and prior to initiating any treatment in the metastatic setting
  Interventions: Genetic: Liquid Biopsy; Genetic: Archival Tumor DNA

INTERVENTIONS:
Genetic: Liquid Biopsy — Patients with metastatic breast cancer in disease progression will undergo a liquid biopsy
Genetic: Archival Tumor DNA — Patients will be prompted to request an archival tumor sample from metastatic origin (preferably) and to send it to the central laboratory for analysis

SUMMARY:
HOPE Focus is an observational study that aims at promoting research against metastatic breast cancer by means of collective research led by patients (patient-centric trial). Patients with metastatic breast cancer living in Spain will voluntarily register and fulfil their journey in the study through the study's digital tool. Mainly they are prompted to answer questionnaires about their disease and expectations, and to provide a blood sample and an archival tumor biopsy. In HOPE Focus these samples will be genomically analyzed and every patient case will be presented in a multidisciplinary molecular advisory board (MAB). The MAB will issue a plain report explaining the significance of the results and will enumerate future therapeutic options that match patient history and his genomic profile, when feasible. Finally, patients will have to answer short follow-up questionnaires twice a year for 3 years.

The study data will allow us to advance implementing precision medicine to improve the management of current and specially future metastatic breast cancer patients.

DETAILED DESCRIPTION:
HOPE Focus - SOLTI-2401 is a prospective, patient-centered research initiative designed to enhance the treatment of patients with MBC through advanced molecular diagnosis in a real-world clinical setting. It uniquely empowers patients to actively participate in their care, from inclusion and data provision to follow-up, utilizing a web-based digital tool (DT) that streamlines their entire journey within the study. The DT not only facilitates seamless communication between patients and the research team, but also serves as a comprehensive repository for relevant study information.

Patients will lead their own inclusion and participation, providing follow-up data through the DT that will guide them during all their journey in the study. After registration and after undergoing an informative interview, eligible patients will provide electronic signature of the informed consent form, and information about their demographic characteristics and relevant oncological information, all through the DT. In addition, the tool will guide them to attend the closest local partner laboratory to:

* Sign a paper version of the informed consent form if it cannot be signed electronically.
* Hand over a tissue block retrieved from their hospital for molecular diagnosis.
* Provide blood for plasma extraction and ctDNA analysis if their disease is progressing to the last line of therapy (liquid biopsy).

The DT will be a reference for patients of the status of their case within the study and will be the main repository of the ICF, clinical information provided by patients, sequencing results and reports generated after Molecular Advisory Board (MAB )discussion. Finally, there will be a three-year active follow-up to capture the impact of molecular diagnosis using the DT.

At the time of disease progression and preferably before the initiation of a new line of therapy, blood will be collected at the closest venue of the partner laboratory. Plasma samples will be tested using a NGS comprehensive panel and a standard genomics report will be generated afterwards.

Participants will be required to provide an archival tumor sample (preferably from a metastatic site) that will undergo genomic characterization. FFPE blocks will be assessed at the study's central laboratory by a pathologist and H&E slides will be digitalized. Samples with sufficient tumor content will undergo DNA extraction, quantification, and quality control. Valid samples will undergo targeted sequencing using a previously validated capture-based panel including more than 400 genes (mutations, CNA) and biomarkers such as tumor mutational burden (TMB) A standard genomic report will be generated after analysis.

Upon genomic report generation (from blood and/or tissue), a SOLTI dedicated team will present the case at the following Molecular Advisory Board (MAB) meeting. During MAB meetings patient cases will be discussed using the new genomic information and the board will issue a report enumerating the potential future therapeutic strategies to be considered.

MAB reports will be in Spanish and will include a text summarizing the interpretation of results. Reports will be addressed to the participants, but they will also be sent to their oncologists (if participating). In addition to the discussion of the molecular results and the treatment recommendations, the MABs are also intended to generate a platform where the HCPs can learn about emerging strategies in MBC management, how to interpret genomics data and embrace fruitful debates to promote continuous learning. The MAB will be gathering a multidisciplinary group of experts in BC clinical management (including medical oncologists and radiation oncologists), cancer geneticists, experts in bioethics, and pathologists. Besides permanent MAB members, physicians treating study participants will be invited to join their patient's discussion.

One month after MAB report delivery, patients will be required to answer a second questionnaire to capture if the information received was relevant for subsequent treatment decisions.

Importantly, the SOLTI-2401 HOPE-Focus Study will not provide any pharmacological intervention to participants. After MAB report delivery, patients will be treated according to local practice or will be directed to ongoing clinical trials. From this moment, patients will be under active follow-up. Periodically, the DT will require them to fill out brief clinical questionnaires to capture the subsequent treatments received. If patients fail to answer a periodic questionnaire, the study team will contact them to reasonably request for response. This follow-up period will last at least 3 years, as SOLTI has the willingness of maintaining the program if the necessary economic supports are achieved, by extending the follow-up period.

Participation of treating physicians will be highly recommended but not mandatory. Patients will be able to request the involvement of their physicians by providing the physician's name and contact details through the web-based digital tool, in accordance with the Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 (GDPR) and the Organic Law 3/2018 on Protection of Personal Data and Guarantee of Digital Rights (LOPDGDD). Only upon electronic written consent collection they will be involved. Then, they will be able to support patient participation and attend the MAB case discussion.

Obtaining patient-reported experience measures (PREMs) of certain aspects involved in cancer care and in molecular diagnosis (knowledge, expectations, concerns, etc.), will allow the design of future strategies to deliver healthcare respecting individual preferences, needs and values. At inclusion and after receiving the report with the MAB assessment, patients will fill out PREM questionnaires. Moreover, during the follow-up process patients will be inquired about their perception of the study's impact on the treatment decisions taken.

The study will be in accordance with the Declaration of Helsinki and Good Clinical Practice Guidelines and applicable regulatory requirements and in accordance with data protection regulations: GDPR and LOPDGDD. Approval of the study protocol will be from an Independent Ethics Committee.

The present initiative intends to build a collaborative patient-centric program for molecular diagnosis in patients with MBC that will facilitate the testing and implementation of novel diagnostic strategies to identify patients who may benefit from precision medicine drugs, either approved or in clinical trials. Moreover, it envisions to promote patient empowerment to live with their disease and to increasing education among HCP and other stakeholders about the potential of molecular diagnosis into MBC care.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients residing in Spain.
2. Age ≥ 18 years.
3. Signed informed consent prior to any study-related procedures, except for registration.
4. Self-reported Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Patients with metastatic breast cancer in at least one of these situations:

   1. Patients recently diagnosed with ER+/HER2- metastatic breast cancer as a recurrence during adjuvant treatment and prior to initiating any treatment in the metastatic setting.
   2. Patients with metastatic breast cancer of any subtype that have progressed after at least one line of treatment in the metastatic setting.

Exclusion Criteria:

1. Presence of a condition or abnormality that, in the opinion of the investigators, would compromise the safety of the patient or the quality of the data.
2. Inability or refusal to commit with the procedures of the study at the moment of inclusion.
3. More than 3 prior systemic chemotherapy or antibody-drug conjugate (ADC) regimens for metastatic disease. Note: treatments for bone metastases (eg, bisphosphonates, denosumab, etc.), targeted therapies (eg, PARP inhibitors, CDK 4/6 inhibitors, immunotherapy etc.) and hormonal therapy are not considered as prior systemic chemotherapy treatments for advanced disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic breast cancer living and being treated in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of incorporating a molecular diagnosis in the management of patients with metastatic breast cancer following a patient-centric strategy. | Ongoing basis during 5 years of study duration
  Percentage of patients with a valid NGS test and a treatment recommendation by the Molecular Advisory Board.

SECONDARY OUTCOMES:
To study the clinical impact of genomic testing in terms of matched therapies prescribed by treating physicians | Ongoing basis during 5 years of study duration
  * Percentage of patients who received a matched therapy against an alteration detected by ctDNA and/or tissue targeted sequencing.
  * Subanalysis based on physician's participation in the study.
Description of Overall Survival (OS) and Progression Free Survival/Time to Next Treatment (PFS/TTNT) of matched treatments. | Ongoing basis during 5 years of study duration
  * Describe PFS/TTNT with treatments directed to molecular targets identified.
  * Describe OS from the moment of registration to the death of the patient.
To study the clinically actionable targets (based on ESCAT) detected using tissue targeted sequencing, and plasma ctDNA targeted sequencing. | Ongoing basis during 5 years of study duration
  Proportion of patients with putatively targetable (ESCAT levels I-II) alterations detected in tissue and plasma ctDNA.
To study the impact of a liquid biopsy based molecular diagnostic in patients with ER+/HER2- BC whose disease progresses as a recurrence during the adjuvant treatment or as a failure of the 1L of treatment or subsequent in the metastatic setting of patie | Ongoing basis during 5 years of study duration
  * ctDNA detection rate in patients with BC whose disease progresses as a recurrence during the adjuvant treatment or as a failure of the 1L of treatment or subsequent in the metastatic setting of patients from any subtype.
  * Frequency of mutations identified in ctDNA, distribution of VAFs and the proportion of patients with a targetable mutation in patients with BC whose disease progresses as a recurrence during the adjuvant treatment or as a failure of the 1L of treatment or subsequent in the metastatic setting of patients from any subtype.
To study the concordance rate for key genomic alterations between ctDNA and tumor targeted sequencing (in a subset of patients who have both samples available). | Ongoing basis during 5 years of study duration
  * Concordance between ctDNA mutation status and tissue mutation status (especially in PI3K-AKT-mTOR pathway genes, ESR1 and HRD and other clinically relevant genes).
  * Concordance between ctDNA and tissue TMB calculations.
To describe the genomic landscape of MBC in a real-world population beyond clinical trials using validated targeted sequencing assays in tissue and ctDNA. Frequency of MBC gene mutations in the study population. | Ongoing basis during 5 years of study duration
  Frequency of MBC gene mutations in the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- SOLTI Cancer Research Group, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided